CLINICAL TRIAL: NCT03036267
Title: Self-care Decision-making: Feasibility of the BREATHE Asthma Intervention Trial
Brief Title: Feasibility of the BREATHE Asthma Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Maureen George, Associate Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AAAR0605
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Asthma Chronic; Health Behavior
Keywords: health disparity; motivational interviewing; African American adults; Federally Qualified Health Centers; adherence; health beliefs; self-management; asthma control
MeSH Terms: conditions — Health Behavior | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE (Experimental): 7-minute brief shared decision-making intervention using a 4-step motivational interviewing approach
  Interventions: Behavioral: BREATHE
- Attention Control Condition (Active Comparator): 7-minute diet and exercise discussion
  Interventions: Other: Attention Control Condition

INTERVENTIONS:
Behavioral: BREATHE — Primary care providers (PCPs) randomized to BREATHE will be trained to deliver the 7-minute brief shared decision-making intervention using a 4-step motivational interviewing approach.
  Other Names: Shared decision-making using motivational interviewing
  Arms: BREATHE
Other: Attention Control Condition — PCPs randomized to the control intervention will not receive any specific training. To control for contact, they will be instructed to engage in a 7-minute diet and exercise discussion as this will not confound results.
  Arms: Attention Control Condition

SUMMARY:
Asthma rates are high and asthma control is greatly reduced in Black, Medicaid-insured adults, due in part to their poor adherence to inhaled corticosteroids (ICS), which in turn may be due to erroneous health beliefs about asthma and negative beliefs regarding ICS. A brief shared decision-making intervention for use by primary care providers in Federally Qualified Health Centers (FQHCs) has the potential to be a novel avenue to greatly improve asthma control in this high-risk patient group.

DETAILED DESCRIPTION:
Uncontrolled asthma disproportionally impacts Black and poor adults. Adherence to inhaled corticosteroids (ICS), which plays a significant role in asthma control, is relatively low in poor and minority populations. Non-adherence to ICS is associated with erroneous personal health beliefs regarding asthma care and with negative beliefs regarding ICS. Despite this, no intervention concurrently addresses beliefs regarding asthma self-care and ICS. Shared decision-making interventions have not been tested in underserved Black adults, despite this model's success in pediatric populations and in White, privately insured patients with asthma. Federally Qualified Health Centers (FQHCs) have unique challenges to helping patients achieve asthma control but are overlooked in asthma intervention research. Process evaluations are often lacking during intervention development. We will address these treatment and methodological gaps.

Objectives: This pilot study will (1) develop a brief shared decision-making intervention delivered by primary care providers (PCPs) to improve asthma control in Black adults receiving care in FQHCs; (2) evaluate the intervention's feasibility and acceptability; and (3) assess preliminary evidence of intervention effects on asthma control, ICS adherence, forced expiratory volume in one second (FEV1) - an objective lung function measure - and asthma quality of life (QOL) over a 3-month follow-up period.

Hypotheses: (1) The intervention will be feasible and acceptable, and (2) over 3 months, relative to controls, patients whose PCPs are trained in the intervention will have significant improvement on asthma control (primary outcome), ICS adherence, FEV1 and asthma QOL (secondary outcomes).

Methods: Using community-based participatory research and including a Patient Advocate, we will develop the intervention, Brief Evaluation of Asthma Therapy (BREATHE). Intervention development is guided by patient and family/support persons of asthma patients input, as well as PCP feedback. We will then conduct a randomized trial of the intervention with 8 PCPs from 2 FQHCs in Philadelphia, PA; for each PCP we will enroll 10 Black adults (N=80) with uncontrolled asthma, and with erroneous asthma care beliefs and negative ICS beliefs. PCPs will be randomized within FQHC to intervention and control; patients will be followed for 3 months. Process evaluation interviews with patients and PCPs will obtain feedback regarding intervention procedures.

Significance: This study has high public health significance because it (1) targets a highly vulnerable population for poor asthma control - Black poor adults with erroneous asthma care beliefs and with negative ICS beliefs; (2) adapts a model-based intervention to develop a novel intervention delivered by PCPs that simultaneously targets erroneous asthma beliefs and negative ICS beliefs, and which has the potential to amplify intervention effects and increase the likelihood of sustainability; and (3) includes a process evaluation, bridging the gap between science and practice, and aiding in the design of a full-scale randomized controlled trial (RCT).

ELIGIBILITY:
The intervention trial will be informed by focus groups

Focus Group Inclusion Criteria:

- Adult patients with persistent asthma or loved ones of adult patients with persistent asthma (prescribed ICS regardless of whether they are using ICS or not) receiving care at the participating FQHCs

Focus Group Exclusion Criteria:

- Patients with persistent asthma or loved ones of patients with persistent asthma under they age of 18 OR NOT prescribed ICS or NOT receiving care at the participating FQHCs

Intervention Inclusion Criteria:

Patients must be:

1. Adults (18 years of age or older)
2. PCP-diagnosed persistent asthma
3. Currently prescribed ICS
4. Receiving asthma care at participating FQHCs
5. Who screen positive for uncontrolled asthma
6. Have erroneous personal health and/or negative ICS beliefs

Intervention Exclusion Criteria:

1. Participation in focus groups during the development phase
2. Non-English speaking
3. Serious mental health conditions (e.g., psychosis) that preclude completion of study procedures or confound analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Spectrum Health Services, Philadelphia, Pennsylvania
  - Greater Philadelphia Health Action, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George M, Arcia A, Chung A, Coleman D, Bruzzese JM. African Americans Want a Focus on Shared Decision-Making in Asthma Adherence Interventions. Patient. 2020 Feb;13(1):71-81. doi: 10.1007/s40271-019-00382-x. PMID 31414396
- [Derived] George M, Pantalon MV, Sommers MLS, Glanz K, Jia H, Chung A, Norful AA, Poghosyan L, Coleman D, Bruzzese JM. Shared decision-making in the BREATHE asthma intervention trial: A research protocol. J Adv Nurs. 2019 Apr;75(4):876-887. doi: 10.1111/jan.13916. Epub 2019 Jan 24. PMID 30479020

RESULTS

PARTICIPANT FLOW:
Groups:
- Focus Groups: Six focus group were held with adults with asthma and their (adult) loved ones
Period: Overall Study
Arm/Group | Focus Groups
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Focus Groups
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 44
  White | 0
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire
Description: Full Title: Asthma Control Questionnaire Construct measured: self-reported asthma control Scoring: 0 points = total asthma control/ best outcome, 6 points = completely uncontrolled asthma/ worst outcome
Time Frame: Baseline - for descriptive purposes only
Population: only those with asthma completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Focus Groups
Number analyzed (Participants) | 32
score on a scale | 2.34 (1.06)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Focus Groups
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03036267/Prot_SAP_000.pdf